CLINICAL TRIAL: NCT02011971
Title: Cognitive Effects of Vinpocetine in Healthy Adults and Patients With Epilepsy
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: We are now considering revision of the IND to determine maximum tolerated dose
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kimford Jay Meador, Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00044949; Stanford Vinpocetine (Other: Other)
Record Dates: First submitted 2013-12-04; First posted 2013-12-16 (Estimated); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy
Keywords: epilepsy; cognition; memory
MeSH Terms: conditions — Epilepsy | interventions — vinpocetine

STUDY DESIGN:
Intervention Model Description: Double-blind single dose crossover with 1-month follow-up open label in patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low dose (Active Comparator): Vinpocetine 10 mg Healthy subjects
  Interventions: Drug: Vinpocetine
- Mid-dose 1 (Active Comparator): Vinpocetine 20mg Healthy subjects
  Interventions: Drug: Vinpocetine
- Placebo (Placebo Comparator): 0 dose of vinpocetine Healthy and Epilepsy subjects
  Interventions: Drug: Vinpocetine
- High Dose (Active Comparator): Vinpocetine 60 mg single dose Healthy Subjects & 20mg tid Epilepsy Subjects
  Interventions: Drug: Vinpocetine

INTERVENTIONS:
Drug: Vinpocetine — Vinpocetine is a chemical obtained from the leaves of the Lesser Periwinkle. It has been shown to improve cerebral metabolism and memory in animals and humans. In addition, it has been shown to enhance long-term potentiation, which has been linked to memory mechanisms. Furthermore, vinpocetine has been shown to have anticonvulsant effects and is more potent than several commonly used antiepileptic drug
  Other Names: ethyl apovincaminate; ethyl apovincaminoate; eburnamenine-14-carboxylic acid ethyl ester; 3 alpha, 16 alpha-apovincaminic acid ethyl ester; ethyl apovincamin-22-oate; Cavinton®; Ceractin; ARGH-4405

SUMMARY:
Pilot studies in healthy volunteers and in patients with epilepsy to assess the potential efficacy and safety of different dosages of vinpocetine in improving cognition.

DETAILED DESCRIPTION:
Cognitive problems are common in patients with epilepsy, but there is currently no specific treatment available. Vinpocetine is a chemical obtained from the leaves of the Lesser Periwinkle. It has been shown to improve cerebral metabolism and memory in animals and humans. In addition, it has been shown to enhance long-term potentiation, which has been linked to memory mechanisms. Furthermore, vinpocetine has been shown to have anticonvulsant effects and is more potent than several commonly used antiepileptic drugs (i.e., carbamazepine, phenytoin, valproate, oxcarbazepine, lamotrigine and topiramate) in inhibiting both sodium and calcium channels, which control release of excitatory neurotransmitters that can lead to brain injury. Thus, vinpocetine might offer a unique drug to help cognition in patients with epilepsy. The investigators propose to conduct pilot studies in healthy volunteers and in patients with epilepsy to assess the potential efficacy and safety of different dosages of vinpocetine in improving cognition.

Specific Aim 1a: To determine if vinpocetine enhances memory and other cognitive functions in healthy volunteers.

Specific Aim 1b: To determine blood levels from 3 different acute oral doses of vinpocetine in healthy volunteers.

Specific Aim 2a: To provide safety and preliminary of efficacy data that vinpocetine can enhance memory and other cognitive functions in patients with epilepsy.

Specific Aim 2b: To determine blood levels from acute and chronic oral doses of vinpocetine in patients with epilepsy as well as effects on anticonvulsant blood levels.

Specific Aim 2c: To provide preliminary of data that vinpocetine can reduce seizure frequency or duration in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria - Healthy (enrollment of healthy volunteers has been completed)

1. Healthy adults 18-60 years old
2. Proficient English
3. Use of appropriate contraception if woman of childbearing potential. This must include complete abstinence for the duration of the study or use of a barrier method plus one other contraceptive method (e.g. hormonal contraception or intrauterine device, IUD).

Inclusion Criteria -Epilepsy

1. Adults (18-60 years old) with localization related epilepsy
2. Patient is on stable antiepileptic drug therapy for last 2 months and is willing to remain on same therapy for the duration of the study.
3. Proficient English
4. Patient complains of memory problems.
5. Neurological Disorders Depression Index -Epilepsy (NDDI-E) score <16
6. Mini-Mental Status Exam (MMSE) score <22
7. No history of status epilepticus in last year
8. No prior epilepsy surgeries
9. Stable antiepileptic drug (AED) therapy for last 2 months or more and willing not to change for 2 months. Vinpocetine will be stopped and the patient will be withdrawn from the study if marked changes occur in seizures or if other adverse events occur.
10. Use of appropriate contraception if woman of childbearing potential. This must include complete abstinence for the duration of the study or use of a barrier method plus one other contraceptive method (e.g. hormonal contraception or IUD).

Exclusion Criteria -Healthy:

1. Major medical disease (e.g., epilepsy, diabetes, heart disease, active cancer, depression)
2. Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening.
3. Use of centrally active medications
4. History of allergy to vinpocetine
5. Scores onintelligence quotient (IQ) <80 or Medical College of Georgia (MCG) Paragraph score < 2 standard deviations below norm.
6. Pregnancy or lactation.

Exclusion Criteria- Epilepsy

1. Major medical disease (e.g., diabetes, heart disease, active cancer, depression)
2. Use of centrally active medications
3. History of allergy to vinpocetine
4. Progressive Cerebral Disease (e.g., Alzheimer's disease)
5. Aphasia
6. Taking more than 3 AEDs
7. Pregnancy or lactation
8. Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the C-SSRS at Screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in CNS Vitals Composite Score | Healthy - weekly treatment visits 1-4; Epilepsy =treatment weeks 4, 8, & 12
  CNS Vitals consists of multiple subtasks that provide an overall composite score will be the primary outcome measure

SECONDARY OUTCOMES:
Adverse Events | Healthy - weekly treatment visits 1-4; Epilepsy =treatment weeks 4, 8, & 12
  safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kimford J Meador, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States